CLINICAL TRIAL: NCT07007169
Title: Mediterranean Diet and Inequality in Early Breast Cancer: A Multicenter Randomized Clinical Trial
Brief Title: Mediterranean Diet and Inequality in Early Breast Cancer
Acronym: MEDITERRACARE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Vejle Hospital (Other); Hospital of Southern Jutland (Other); Odense University Hospital (Other); Syddansk Universitet, Denmark (Unknown); University of Copenhagen (Other); Aarhus University Hospital (Other); Danish Breast Cancer Cooperative Group (Other); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 629752-24 S-20240087
Record Dates: First submitted 2025-03-31; First posted 2025-06-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Early Breast Cancer
Keywords: Microbiome; Mediterranean Diet; Inequality in cancer; Chemotherapy; Adjuvant; Neoadjuvant; Short-chain Fatty Acids
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized 2:1 to Mediterranean Diet versus standard diet; controlled; blinding is not possible
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Experimental): The intervention is the Mediterranean Diet.
  Interventions: Dietary Supplement: The goal is daily consumption of a minimum of 30 grams of dietary fiber and weekly consumption of a minimum of 30 different plant foods; minimizing the amount of ultra-processed food.
- Standard Diet (Active Comparator): The control group will continue their normal diet.
  Interventions: Other: Standard Diet

INTERVENTIONS:
Dietary Supplement: The goal is daily consumption of a minimum of 30 grams of dietary fiber and weekly consumption of a minimum of 30 different plant foods; minimizing the amount of ultra-processed food. — The intervention group will receive personalized education and guidance from a nutrition therapist.
  Arms: Mediterranean Diet
Other: Standard Diet — The control group will continue their normal diet, and not receive guidance or participate in group sessions.
  Arms: Standard Diet

SUMMARY:
Social determinants such as education, income, marital status, and social networks play a crucial role in cancer outcomes, including breast cancer. One potential influencing factor is diet, and the Mediterranean diet has been shown to benefit both the health and the microbiome.

This raises the question: Does adherence to the Mediterranean diet impact the microbiome, quality of life, overall well-being, and outcomes in breast cancer patients undergoing (neo)adjuvant treatment, particularly among those with unfavorable socioeconomic determinants?

The Mediterranean diet consists of plant foods such as vegetables, fruits, nuts, seeds, berries, legumes, herbs, and spices. It also features animal proteins like fish, meat, and cheese, along with fat from olive oil. Thus, adherence to the Mediterranean diet is adherence to the official Danish diet recommendations.

This phase II clinical trial is an interdisciplinary study combining nutrition, sociology, and health research. Breast cancer patients candidates for (neo)adjuvant treatment at four oncology departments in Region South Denmark will be randomized 2:1 to the Mediterranean diet (with individual dietary guidance from a nutrition therapist aiming at daily consumption of a minimum of 30 grams of dietary fiber and weekly consumption of a minimum of 30 different plant foods; minimizing the amount of ultra-processed food) versus the patient's regular diet, in conjuction with the (neo)adjuvant chemotherapy.

The trial's primary endpoint will be changes in gut microbiota composition in feces.

The study evaluates how the Mediterranean diet affects the microbiota (evaluated using Oxford Nanopore Technology 16S sequencing on fecal samples); short-chain fatty acids in stool and plasma (assessed by mass spectrometry); immune system (using flow cytometry for immune cell determination in blood and immunohistochemical determination of immune cells in the tumor tissue); and patients' social quality of life, overall well-being, sense of empowerment, and personal feeling of agency (using the WHOQOL-100 questionnaire); taking into account the impact of the distance from the patient residence to the hospital (tracked from GEOTEAM at Statistics Denmark), and socioeconomic factors (using the DREAM database).

The evaluation of biological parameters is based on the suggested mechanism of action. A diet rich in various plant foods and dietary fiber will alter the gut microbiota, promoting bacteria producing high amounts of short-chain fatty acids. These fatty acids will activate immune cells, aiding in the destruction of cancer cells.

The study will also assess whether the Mediterranean diet will positively impact the patients' social quality of life, overall well-being, sense of empowerment, and personal feeling of agency. The Mediterranean diet may not only lead to improved dietary habits but also serve as a crucial tool for breast cancer patients, particularly among those with unfavorable socioeconomic determinants. Enhanced empowerment and improved coping tools could be an important step in combating cancer-related inequalities.

DETAILED DESCRIPTION:
STUDY PURPOSE The project investigates whether adherence to the Mediterranean diet can influence the microbiome, improve quality of life, overall well-being, sense of empowerment, personal feeling of agency, immune activity, levels of short-chain fatty acids and patient outcomes in breast cancer patients undergoing chemotherapy. Additionally, it examines if these effects are more pronounced in individuals with challenging socioeconomic determinants.

BREAST CANCER Among women, breast cancer is the most diagnosed cancer, and is the leading cause of cancer deaths globally in most countries, with 2.3 million new cases recorded in 2022 and approximately 665,000 deaths. In Denmark, there are 5000 new cases, and 1.050 deaths annually, of those 250 in the Region of Southern Denmark. In men, breast cancer is rare with an average of 42 new cases annually in Denmark.

ONCOLOGICAL TREATMENT The oncological treatment of early breast cancer encompasses neoadjuvant (pre-surgery) and adjuvant (post-surgery) treatments.Chemotherapy comprising anthracyclines and taxanes is a cornerstone in both neoadjuvant and adjuvant settings for breast cancer treatment. These drugs have been shown to significantly improve patient outcomes as these regimens are particularly effective in shrinking tumors before surgery, reducing the risk of recurrence and improving overall survival. HER2-targeted therapies, such as trastuzumab, are specifically used for HER2-positive breast cancers in conjunction with chemotherapy and have significantly improved outcomes. Recently, checkpoint immunotherapy, pembrolizumab, has been approved in Denmark for triple-negative early breast cancer together with chemotherapy due to increased pathological complete response (pCR).

SOCIOECONIC INEQUALITY At the national level, disparities in breast cancer outcomes are commonly observed along socioeconomic and demographic lines in both low-, middle- and, high-income countries. These disparities are evident across all stages of the breast cancer continuum, from exposure to modifiable risk factors to access to palliative care and mortality rates. Consequently, women with lower socioeconomic status are more likely to present with late-stage cancer and experience poorer breast cancer prognoses compared to those with higher socioeconomic status. Cancer inequalities at the individual level are predominantly shaped by systemic social determinants of health.

In Denmark an estimated 21% of breast cancer deaths five years after the diagnosis of breast cancer could have been avoided, had patients in all income groups had the same survival rate as the high-income group. Thus, social inequality in cancer survival is a critical problem, and patients with little education, low income, or living alone have poorer survival than better educated cancer patients, with higher income, and living in a relationship. This applies despite women with higher socioeconomic status having significantly higher breast cancer incidence.

GUT MICROBIOTA AND MEDITERRANEAN DIET The human gut hosts approximately 38 trillion cells called the microbiota; the human gut microbiome consists of the genes these cells harbor.

In the 2022 update of Hallmarks of Cancer, the microbiome was introduced as a new important hallmark of cancer. Importantly, the microbiome modulates four other hallmarks: tumor growth, tumor-promoting inflammation, immune evasions, and genomic instability; additionally, the microbiome modulates therapy resistance. The implication is, therefore, that the microbiome is a critical link in cancer development, progression, and treatment response.

The Mediterranean diet is defined as the consumption of fresh fruits, vegetables, nuts, berries, legumes, and non-refined cereals. Olive oil is the principal source of lipids. Moderate intake of alcohol, preferably red wine, with meals; moderate consumption of fish, poultry, eggs, low-fat dairy products, and sweets; monthly consumption of red meat; and regular physical activity.

As the Mediterranean diet includes a wide variety of plant foods and proteins from animal sources, it is a flexible option for many patients. It is not restrictive and allows for many different types of food, with the main limitation being processed foods. This flexibility was a key reason why Harvey et al. chose this diet for a randomized clinical trial involving cancer patients. The study aimed to measure fatigue during chemotherapy and included a sub-study to qualitatively assess how patients felt about making dietary changes during their treatment, identifying facilitators and barriers. Importantly, patients reported that the diet gave them a sense of control and empowerment. They enjoyed learning about nutrition, trying new foods, feeling in control, setting goals, doing something constructive to aid their treatment, and having a positive focus. Barriers included chemotherapy side effects (mouth sores, taste changes, and lack of energy) and food preferences.

Higher adherence to the Mediterranean diet was associated with a 23% lower risk of all-cause mortality. The Mediterranean diet was feasible and safe for adults with cancer. Mediterranean diet has been associated with a reduced risk of breast cancer development. Its impact on survival outcomes after breast cancer diagnosis remains an area of active investigation. Changes in the microbiome composition were observed already after four weeks of the Mediterranean diet.

The Mediterranean diet has several effects, including lipid-lowering and anti-inflammatory actions, reducing chronic inflammation. Moreover, bacteria in the gut ferment dietary fiber to short-chain fatty acids; factors that upregulate immune functions. Short-chain fatty acids are important as an energy source for intestinal epithelial cells, but some enter the bloodstream and act as signaling molecules. They target G-protein-coupled receptors (GPCR) GPCR41, GPCR43, and GPCR109A.

Several studies in patients with melanoma, and cancers of the kidney, lung, and bladder have found that bacterial diversity at baseline can predict response to immunotherapy treatment; some types of bacteria are often reported to be found in larger quantities at baseline in responders than in non-responders, especially Akkermansia mucinifila, Ruminococcaceae, Faecalibacterium, and Lachnospiraceae.

In patients with primary HER2-positive breast cancer undergoing trastuzumab treatment, a recent study revealed the direct involvement of the gut microbiota in trastuzumab efficacy. To the extend of our knowledge, the association with response to checkpoint immunotherapy in breast cancer patients has not been reported.

MICROBIOME AND VITAMIN D Vitamin D has recently been associated with changes in the microbiome and cancer outcomes. Vitamin D is the only vitamin not normally consumed sufficiently even in a well-balanced diet. The main source of vitamin D is solar exposure to the skin. Denmark is situated between the 55th and 57th northern latitudes and therefore UV exposure is insufficient for vitamin D production for large parts of the year. Measurements of vitamin D will be performed at baseline and at Day 1 of cycle 6, and daily supplementation with 50 micrograms of vitamin D is encouraged.

POTENTIAL BENEFITS AND RISKS The potential benefits are that the Mediterranean diet will result in greater microbial diversity during (neo)adjuvant therapy, increase the amounts of short-chain fatty acids in serum and stool, activate the immune system, and improve patient outcomes.

Moreover, the Mediterranean diet may positively impact the patient's social quality of life, overall well-being, sense of empowerment, and personal feeling of agency.

Additionally, these effects may be more pronounced in individuals with challenging socioeconomic determinants.

The potential risk of harm is considered minimal since the intervention is food, and the investigated Mediterranean Diet is comparable to the diet recommended by the Danish Health Authorities (foedevarestyrelsen.dk) The study will be carried out according to the principles outlined in the Declaration of Helsinki. With food as the intervention, the study does not need monitoring from the GCP unit, according to Danish rules.

INTERVENTION The intervention is the Mediterranean Diet.

STUDY POPULATION The study population consists of patients with newly diagnosed early breast cancer, candidates for (neo)adjuvant chemotherapy-based treatment at one of the participating sites in the Region of Southern Denmark.

PATIENT INVOLVEMENT A patient panel, comprising four breast cancer survivors and one representative from a cancer patient association, is actively involved in the design and execution of the MEDITERRACARE study helping developping patient information material, review and provide feedback on questionnaires, and offer practical insights for conducting the trial.

RELEVANCE OF THE TRIAL Changes in bacterial composition can occur within a few weeks of switching to a diet rich in dietary fiber and various plant foods. A positive correlation between gut microbiota and favorable outcomes to checkpoint immunotherapy has been demonstrated in cancer patients. Gut microbiota is important for HER2+ therapy efficacy.

Socioeconomic inequalities are critical for breast cancer patients. The study will evaluate whether adherence to the Mediterranean diet can influence the microbiome, and improve quality of life, overall well-being, sense of empowerment, personal feeling of agency, immune activity, amounts of short-chain fatty acids, and patient outcomes in breast cancer patients undergoing chemotherapy. Additionally, it examines if these effects are more pronounced in individuals with challenging socioeconomic determinants.

This study addresses a knowledge gap. No study worldwide has assessed the Mediterranean diet in early breast cancer patients during chemotherapy with special emphasis on socioeconomic inequality.

HYPOTHESIS The hypothesis is that the Mediterranean diet results in greater microbial diversity during (neo)adjuvant therapy, increases the amounts of short-chain fatty acids in serum and stool, increases the numbers of T- and Natural Killer cells in blood and tumor tissue, reduces inflammation in blood and tumor tissue, and improves patient outcomes.

Moreover, the Mediterranean diet will positively impact the patient's social quality of life, overall well-being, sense of empowerment, and personal feeling of agency.

Additionally, these effects will be more pronounced in individuals with challenging socioeconomic determinants.

STUDY DESIGN The MEDITERRACARE study is designed as a phase II randomized, controlled trial with two arms in a 2:1 allocation ratio evaluating the Mediterranean diet versus regular diet, and a primary endpoint of changes in gut microbiota composition. The study protocol is reported following the CONSORT guidelines.

STUDY SETTING AND RECRUITEMENT Enrolment takes place at four Danish oncology outpatient clinics in the Region of Southern Denmark (Odense, Vejle, Sønderborg, Esbjerg).

Randomization will be performed as block randomization with 2:1 allocation using a computer-generated table of block sizes of 6 or 9, created and supervised by a data manager at OPEN, Open Patient Data Explorative Network, Odense University Hospital, Region of Southern Denmark.

Blinding of patients and health care professionals involved is not intended.

DETAILS ON INTERVENTION The patients randomized to the intervention arm, and if possible a partner or other family member, will receive nutritional guidance during the weekly outpatient chemotherapy visits or via online calls or home visits. Initially 1x weekly during the first month and every other week onwards. In addition, patients will get a booklet on how to implement the Mediterranean Diet in daily life, and access to a password-protected website with teaching videos and Mediterranean diet recipes. To ensure compliance regarding sampling of feces and reporting of food intake patients in the control arm will also be called on during visits to the department.

Group sessions will be arranged for patients randomized to the Mediterranean diet and a hot-line is open during working hours.

DATA COLLECTION Study data will be collected and managed using the REDCap electronic data capture tool (Vanderbilt University, v.12.0.33) hosted at OPEN (Open Patient Data Explorative Network, Odense University Hospital).

At the first consultation at the Department of Oncology, a blood test will be drawn for baseline values and kits for stool sampling at home will be provided to the patient. The stool sample should be obtained at home before the chemotherapy starts.

TIMING DATA COLLECTION The WHOQOL-100 questionnaire and baseline dietary and lifestyle questionnaire will be provided to the patient's E-boks. Data will be captured in REDCap.

Stool samples (1-2 grams per collection) will be collected by patients at home and immediately frozen at -18°C in their home freezer. Patients will bring their samples to the hospital in a cooling bag at the next planned visit and the samples will immediately be transferred to -20°C until DNA extraction. Stool samples will be obtained at baseline, and at Day 1 of cycle 2, 4, 6, or in case of early discontinuation of chemotherapy and stored in a research biobank until completion of primary analyses. Potential left-over stool or Bacterial DNA after the analyses for this study are stored in the OPEN BIOBANK for future, not yet specified, research. Participants will be contacted and asked for consent in case of future research.

Microbiome evaluation will use Oxford Nanopore Technology 16S sequencing of fecal samples.

Metabolome assessment will detect short-chain fatty acids (SCFAs) in patient stool and plasma samples using ultrahigh-performance liquid chromatography-tandem mass spectrometry.

Adhesion to the diet will be measured via food diaries (www.myfood24.org). The software provides feedback to the user about reaching the daily/weekly goals, thereby nudging the participant to reach the target. Patients will also fill out a paper record of different plant foods eaten every week.

Quantification of CD4+ T-cells, CD8+ T-cells, CD19+ B cells, and 56+ Natural Killer cells will be performed by flow cytometry.

Hematology (hemoglobin, white blood cell count, absolute neutrophils, monocytes, lymphocytes, and platelet count) CRP, Vitamin D status will be measured at initiation of the study and at day 1 of chemotherapy cycle 6.

GlycA and lipoproteins will be examined using Nuclear Magnetic Resonance (NMR)-technique at Nightingale, Finland, (https://nightingalehealth.com) as an expression of metabolic improvements.

Blood samples drawn after a minimum of 6 hours fasting will be treated and stored according to current research ethical practice in Denmark in a research biobank assigned for this trial. Blood samples of a total of 40 ml/time are drawn at four time points: at baseline, and Day 1 of cycle 2, 4, and 6 chemotherapy, or in case of early discontinuation of chemotherapy.

Samples are stored as plasma, serum, buffy coat, and whole blood at minus 80 degrees Celsius at the Departments of Biochemistry of participating hospitals and final storage at the OPEN BIOBANK and stored in a research biobank until completion of primary analyses. Potential left-over blood after the analyses for this study are stored in the OPEN BIOBANK for future, not yet specified, research. Participants will be contacted and asked for consent in case of future research.

Archived tumor tissue from the primary breast tumor will be sampled, including the diagnostic biopsy and surgery specimens in neoadjuvant-treated patients, and the surgery specimens in adjuvant-treated patients, which are then stored in a research biobank. Primary tumor tissue will be analyzed for tumor-infiltrating immune cells.

Pathological samples are stored according to clinical routines at the Departments of Pathology affiliated with the trial sites. Immunohistochemical staining will be performed at the Department of Pathology, Esbjerg Hospital.

The following immune cells will be identified within the tumor tissue: CD8+ T cells, CD4+ T cells, FoxP3 regulatory T Cells, CD20+ B Cells, CD57+ NK Cells, CD66b+ Neutrophils granulocytes, CD68+ Macrophages, Granzyme B (GZMB)+ Cells, PD-L1. These immune cells will be quantified using digital image analysis combined with artificial intelligence at the Department of Clinical Medicine, Aarhus University. The median cell density of immune cells per mm2 tumor tissue will be calculated.

DATA REGISTRATION Data will be collected in a secure and central REDCap database. Groups and subgroups Participating patients should have newly diagnosed early breast cancer and be considered eligible for initiating either adjuvant or neoadjuvant chemotherapy-based treatment.

DURATION OF PARTICIPATION In MEDITERRACARE, patients will be followed from randomization before chemotherapy commencement until the start of treatment cycle 6. If a patient stops chemotherapy before cycle 6, blood and fecal samples are collected and participation in the trial ends. Recruitment is planned to begin uniformly across centers from April 2025. The recruitment period is expected to last 18 months.

Data collection is planned to cease latest April 2027, with primary study reporting completed by April, 2028. Follow-up for clinical events, i.e. recurrence, will be conducted through Danish Breast Cancer Cooperative Group(DBCG) database until December 2036. Follow up for for vital status will be followed up via the Central Person Register (CPR) registry until December 2036.

STOPPING THE TRIAL The sponsor can stop the trial in case of practical issues such as insufficient inclusion of patients.

RANDOMIZATION CODE The randomization code will be stored in the REDCap database. Code breaking is not relevant in the MEDITERRACARE study.

CASE REPORT FILES (CRFs) Data to be extracted from the hospital records will be directly typed into the central REDCap database.

Questionnaires filled out by the patient electronically at home will directly be stored in the central REDCap database. Questionnaires filled out by the patient on paper (plants consumed per week) will be collected and typed into the REDCap database.

Patients can stop participating in the trial at any time point without explanation.

EXCLUSION OF GENDER OR AGE GROUPS There are no restrictions on age and gender except for restricting the participation to adults. Breast cancer is extremely rare below the age of 18.

As breast cancer is rare in males, we expect only a few males to be recruited. As the oncology department typically handles breast cancer in males, we do not expect males to be underrepresented.

SOCIOECONOMIC EQUALITY AND PATIENT QUALITY OF LIFE The driving question in this part of the study is whether the Mediterranean diet will positively impact the patients' social quality of life, overall well-being, sense of empowerment, and personal feeling of agency, using the WHOQOL-100 questionnaire.

We will explore both geographic and social inequality, based on our previous extensive research in this area encompassing both geographic and social inequality in health.

The distance to the healthcare system is defined as the geographical distance between the patient's place of residence and the hospital. The distance calculation is carried out by GEOTEAM at Statistics Denmark.

Co-variables include socio-demographic and socio-economic characteristics, such as age, gender, cohabitation status, employment, income, and education, in addition to disease stage and co-morbidity. These will be obtained from relevant registers in the DREAM database, such as income, education, and employment.

In the qualitative study, the focus is on the experience of the intervention, and the benefits or barriers associated with it. The emphasis is on patients' everyday experiences, how the intervention affects their practical lives, and whether they encounter challenges and, if so, what those challenges are. The qualitative interview study is based on semi-structured interviews with 20 patients, of whom 15 have received the Mediterranean diet intervention and 5 have not.

First, the register analysis will be performed to establish a foundational understanding of the participants' socio-economic and socio-demographic conditions. Second, responses from utilizing the WHOQOL-100 questionnaire will analyzed. Third, individual interviews will be conducted with the patient group, focusing on uncovering their experiences, practices, and perspectives regarding their life situations and overall well-being. Moreover, data on family/relatives support on dietary changes and support in general for women under critical risk will be extracted.

ADHERENCE Adherence to the protocol will be monitored via food registration in the MyFood24 system. Patients are required to report their daily food intake at least 3 days per week. Every week a separate report on weekly intake of different plants should be filled out.

Patients are required to fill out the forms, and will be encouraged to fulfill the goals of consuming 30 grams of dietary fiber daily and 30 different plants per week in the intervention group and follow their normal diet in the control group.

COMPLIANCE AND MONITORING Compliance will be monitored via MyFood24 and by collection of plant registration forms.

SUBSEQUENT TREATMENT If a patient leaves the trial, they will continue their normal medical treatment without the diet intervention.

SAFETY EVALUATION Since the MEDITERRACARE study is a clinical trial investigating a diet similar to that recommended by the Danish Health Authorities, there will be no safety issues to assess.

STATISTICS Data will be stored in a secure server in OPEN Analysis. Descriptive analyses will be performed to explore exchangeability between the two study arms and presented in a table describing the study population on key characteristics.

The WHOQOL-100 questionnaire will be analyzed. A DREAM database analysis will be performed to establish an understanding of participant's socioeconomic and socio-demographic levels. Individual interviews will be conducted to uncover experiences, practices, and perspectives regarding their life situation and general well-being.

The analysis will separate participants into three socio-economic groups (low-risk vs. median-risk vs. high-risk). This stratification will be used as the key to interpreting data for gut bacteria composition and immune cell activity For comparison between groups two-sample Student's t-test will be applied for normally distributed numerical data and the Wilcoxon-Mann-Whitney test will be applied for non-normally distributed numerical data while categorical data will be compared by chi-squared test.

Correlation analyses of median values (measured at the start of cycle 6) of the six domains in the WHO-100 questionnaire, and median estimates (measured at the start of cycle 6) of blood CRP, monocytes, neutrophils, CD4/CD8/CD19/CD56 cells as well as median values of daily dietary fiber and median weekly plant food intake; concentrations of fecal metabolites including SCFA, and alpha diversity, beta diversity as well as microbial differential abundance will be performed with relevant stats package within the statistical programming language R (v.3.5.1).

A recurrence will be defined as any invasive breast cancer recurrence irrespective of localization.

Information on overall survival will be retrieved by linkage to the national CPR registry.

Invasive disease-free survival among groups will be analyzed in crude analysis using the Kaplan-Meier and distant recurrence-free survival will be analyzed using competing risk analysis with cumulative incidences. Cox regression hazards analysis will be performed allowing for controlling for confounders in multivariable analysis.

A 2-sided p-value of ≤ 0.05 will be used to determine significance. All statistical data analysis will be carried out using R.

SAMPLE SIZE CONSIDERATIONS Assuming a larger heterogeneity in the intervention group of a factor of sqrt(2) (due to compliance and the dietary flexibility for the intervention) and with a distribution of 2:1 between intervention and standard diet, the relative effect size detectable on the change from baseline to the end of intervention should be 0.69 with n = 33 in the standard diet group and n = 66 in the intervention group to have a study power of 0.8 with a significance level of 0.05. Thus, assuming a 5% drop-off, the study needs 105 patients to be included. There will be stratification for neoadjuvant chemotherapy versus adjuvant chemotherapy.

INTERIM ANALYSIS IS NOT PLANNED Missing data will be handled according to the scoring instructions of the instruments or imputations.

Deviations from the statistical analysis plan will be reported in the final publications.

All analyses will be performed as intention-to-treat analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent approved by the Ethical Review Board.
2. Age ≥ 18
3. Histologically confirmed unilateral adenocarcinoma of the breast, stage I-III, candidates for neoadjuvant chemotherapy followed by curative surgery, or adjuvant chemotherapy after curative surgery, according to the Danish Breast Cancer Group guidelines 48. The addition of trastuzumab and pertuzumab in HER2-positive tumors, or pembrolizumab in triple-negative tumors, per Danish Breast Cancer Group guidelines 48, is allowed as an adjunct to chemotherapy.
4. Good performance status (WHO performance status 0 or 1).
5. Willingness by the patient to undergo treatment and study-related procedures according to the protocol.
6. Have a smartphone or computer to which it is possible to receive emails (for food diary; www.myfood24.org)
7. Must be willing to restrict from probiotic (living microorganisms) supplements during the study. Fermented foods are allowed.

   -

Exclusion Criteria:

1. Clinical or radiological signs of metastatic disease.
2. History of other malignancy within the last 5 years, except for carcinoma in situ of the cervix or non-melanoma skin cancer.
3. Previous chemotherapy for cancer or other malignant disease.
4. Major altered digestive system disorders (e.g. gastric by-pass or Crohn's disease or ulcerative colitis)
5. Unable to communicate effectively in Danish or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Change in microbiota composition | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  The primary objective of this trial, assessing the clinical efficacy of the Mediterranean diet, is changes in gut microbiota composition, analyzed as microbial differential abundance (measures the difference in the abundance of specific microbial taxa between groups) by the ZicoSeq differential abundance analysis method, accounting for multiple-testing using the false discovery method (FDR). The endpoint will be measured at cycle 6 and compared with baseline values, in patients allocated to the Mediterranean Diet compared to patients on their regular diet.

SECONDARY OUTCOMES:
Change in alpha diversity in stool samples | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Alpha diversity in stool samples, at Day 1 of chemotherapy cycle 2, 4, or 6, compared with baseline values, in the Mediterranean diet group compared to the regular diet group, to evaluate species richness and evenness within each sample. Alpha diversity will be assessed using the Shannon diversity index and tested using paired t-test.
Change in beta diversity in stool samples | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Beta diversity in stool samples, at Day 1 of chemotherapy cycle 2, 4, or 6, compared with baseline values, in the Mediterranean diet group compared to the regular diet group, visualizing the differences in microbial communities between samples. Beta diversity will be assessed using Bray-Curtis dissimilarity metrics followed by Principal Coordinates Analysis for visualization and permanova for statistical inference
Level of short-chain fatty acids in stool and plasma | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of short-chain fatty acids in stool and plasma, at Day 1 of chemotherapy cycle 2, 4, or 6, compared with baseline values, in the Mediterranean diet group compared to the regular diet group.
Quality of life measured by WHOQOL-questionnaire | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Quality of life, overall well-being, and the sense of agency, at Day 1 of chemotherapy cycle 2, 4, or 6, compared with baseline values, in the Mediterranean diet group compared to the regular diet group, evaluated by the World Health Organisation Quality of Life (WHOQOL)-100 questionnaire, a comprehensive tool developed by the World Health Organization to assess various aspects of quality of life (QOL) and translated into Danish. It consists of 100 questions that cover six broad domains: physical health, psychological health, level of independence, social relationships, environment, and spirituality/religion/personal beliefs. Responses are recorded on a 5-point Likert scale, where 1 is the worst score and 5 is the best score. The mean score will be calculated for each domain and facet, with higher scores indicating a better quality of life.
Socioeconomic factors and quality of life correlated with microbiome composition and diversity | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of education, income, marital status, social networks, and quality of life World Health Organisation Quality of Life (WHOQOL-100) correlated with microbial differential abundance, alpha diversity, and beta diversity in the Mediterranean diet cohort compared with the standard diet cohort.
Invasive disease-free survival (IDFS) | From enrollment in study and follow up for 10 years.
  Invasive disease-free survival (IDFS), defined as the time from randomization until the date of the first occurrence of one of the following events:
  * Ipsilateral invasive breast tumor recurrence: invasive breast cancer involving the same breast parenchyma as the original primary.
  * Regional invasive breast cancer recurrence: Invasive breast cancer in the axilla, regional lymph nodes, chest wall, and skin of the ipsilateral breast.
  * Distant recurrence: Metastatic disease-breast cancer that has either been biopsy confirmed or clinically diagnosed as recurrent invasive breast cancer.
  * Death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
  * Contralateral invasive breast cancer.
  * Second primary non-breast invasive cancer
Distant recurrence-free survival | From enrollment in study and follow up for 10 years.
  Distant recurrence-free survival, defined as the time from randomization to first occurrence of distant recurrence, or death of any cause, with loco-regional recurrence, contralateral breast cancer and second primary non-breast invasive cancer competing events.
Overall survival (OS) | From enrollment in study and follow up for 10 years.
  Overall survival, defined as the time from randomization to death attributable to any cause, including breast cancer, non-breast cancer, or unknown cause.
Rate of pathological response | Baseline to date of surgery in neoadjuvant patients.
  Rate of pathological response (only in patients on neoadjuvant therapy).

OTHER OUTCOMES:
Level of CD4+ T-cell immune activity in blood | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of immune activity, measured as the number of blood CD4+ T-cells from baseline to Day 1 of chemotherapy cycle 2, 4, or 6, in the two diet arms.
Level of CD8+ T-cell immune activity in blood | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of immune activity, measured as the number of blood CD8+ T-cells from baseline to Day 1 of chemotherapy cycle 2, 4, or 6, in the two diet arms.
Level of CD 56+ Natural Killer cell immune activity in blood | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of immune activity, measured as the number of blood CD4+ T-cells, CD8+ T-cells, or CD56+ Natural Killer cells from baseline to Day 1 of chemotherapy cycle 2, 4, or 6, in the two diet arms.
Level of CD8+ T-cell immune activity from baseline biopsy to definite surgery | Baseline to date of surgery in neoadjuvant patients.
  Level of immune activity, measured as the number of tumor-infiltrating CD8+ T-cells from baseline biopsy to definite surgery in patients on neoadjuvant therapy, in the two diet arms.
Level of CD57+ NK cell immune activity from baseline biopsy to definite surgery | Baseline to date of surgery in neoadjuvant patients.
  Level of immune activity, measured as the number of tumor-infiltrating CD57+ Natural Killer cells from baseline biopsy to definite surgery in patients on neoadjuvant therapy, in the two diet arms.
Level of neutrophil immune activity from baseline biopsy to definite surgery | Baseline to date of surgery in neoadjuvant patients.
  Level of immune activity, measured as the number of tumor-infiltrating neutrophils from baseline biopsy to definite surgery in patients on neoadjuvant therapy, in the two diet arms.
Level of inflammation marker (blood neutrophils) | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of inflammation (blood neutrophils) from baseline to Day 1 of chemotherapy cycle 2, 4, or 6, in the two diet arms.
Level of inflammation marker (monocytes) | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of inflammation (monocytes) from baseline to Day 1 of chemotherapy cycle 2, 4, or 6, in the two diet arms.
Level of inflammation marker (CRP) | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of inflammation (C-reactive protein (CRP)) from baseline to Day 1 of chemotherapy cycle 2, 4, or 6, in the two diet arms.
Level of inflammation marker (neutrophil/lymphocyte ratio) | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of inflammation (neutrophil/lymphocyte ratio) from baseline to Day 1 of chemotherapy cycle 2, 4, or 6, in the two diet arms.
Degree of adherence to dietary intervention | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision, as per clinician decision.
  The degree of adherence to the dietary intervention, measured as a percentage of patients reaching the goal of 30 plants per week and 30 grams of fiber daily.
Qualitative interview on facilitators and barriers to adherence to dietary intervention | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Facilitators and barriers to adherence to dietary intervention during chemotherapy treatment, assessed by qualitative interviews
Level of GlycA in blood | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of GlycA from baseline to Day 1 of chemotherapy cycle 2, 4, or 6 in the two diet arms.
Level of vitamin D in blood | Baseline to start of cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of vitamin D from baseline to Day 1 of chemotherapy cycle 6 in the two diet arms.
Level of lipoproteins in blood | Baseline to Day 1 of chemotherapy cycle 6. Each cycle is 3 weeks for regular schedule or 2 weeks for accelerated schedule, as per clinician decision.
  Level of lipoproteins from baseline to Day 1 of chemotherapy cycle 2, 4, or 6 in the two diet arms.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - University Hospital of Southern Denmark, Esbjerg, Esbjerg
  - Sygehus Lillebaelt, Vejle, Vejle

IPD SHARING:
Plan to Share IPD: Yes
When the clinical trial ends, the anonymized data will be made available to other researchers through public databases such as the Zenodo open data repository (CERN) or other equivalent databases.
Supporting Information: Study Protocol
Time Frame: when the clinical trial ends and data are mature, anticipated 1 January 2031
Access Criteria: Zenodo open data repository (CERN) or other equivalent databases.

REFERENCES:
- [Background] Spencer CN, McQuade JL, Gopalakrishnan V, McCulloch JA, Vetizou M, Cogdill AP, Khan MAW, Zhang X, White MG, Peterson CB, Wong MC, Morad G, Rodgers T, Badger JH, Helmink BA, Andrews MC, Rodrigues RR, Morgun A, Kim YS, Roszik J, Hoffman KL, Zheng J, Zhou Y, Medik YB, Kahn LM, Johnson S, Hudgens CW, Wani K, Gaudreau PO, Harris AL, Jamal MA, Baruch EN, Perez-Guijarro E, Day CP, Merlino G, Pazdrak B, Lochmann BS, Szczepaniak-Sloane RA, Arora R, Anderson J, Zobniw CM, Posada E, Sirmans E, Simon J, Haydu LE, Burton EM, Wang L, Dang M, Clise-Dwyer K, Schneider S, Chapman T, Anang NAS, Duncan S, Toker J, Malke JC, Glitza IC, Amaria RN, Tawbi HA, Diab A, Wong MK, Patel SP, Woodman SE, Davies MA, Ross MI, Gershenwald JE, Lee JE, Hwu P, Jensen V, Samuels Y, Straussman R, Ajami NJ, Nelson KC, Nezi L, Petrosino JF, Futreal PA, Lazar AJ, Hu J, Jenq RR, Tetzlaff MT, Yan Y, Garrett WS, Huttenhower C, Sharma P, Watowich SS, Allison JP, Cohen L, Trinchieri G, Daniel CR, Wargo JA. Dietary fiber and probiotics influence the gut microbiome and melanoma immunotherapy response. Science. 2021 Dec 24;374(6575):1632-1640. doi: 10.1126/science.aaz7015. Epub 2021 Dec 23. PMID 34941392
- [Background] Tanggaard Andersen P, Holst Algren M, Fromsejer Heiberg R, Joshi R, Kronborg Bak C. Social network resources and self-rated health in a deprived Danish neighborhood. Health Promot Int. 2018 Dec 1;33(6):999-1009. doi: 10.1093/heapro/dax051. PMID 28973140
- [Background] Kim KS, Lee Y, Chae W, Cho JY. An Improved Method to Quantify Short-Chain Fatty Acids in Biological Samples Using Gas Chromatography-Mass Spectrometry. Metabolites. 2022 Jun 7;12(6):525. doi: 10.3390/metabo12060525. PMID 35736458
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Mandal S, Van Treuren W, White RA, Eggesbo M, Knight R, Peddada SD. Analysis of composition of microbiomes: a novel method for studying microbial composition. Microb Ecol Health Dis. 2015 May 29;26:27663. doi: 10.3402/mehd.v26.27663. eCollection 2015. PMID 26028277
- [Background] Yang L, Chen J. A comprehensive evaluation of microbial differential abundance analysis methods: current status and potential solutions. Microbiome. 2022 Aug 19;10(1):130. doi: 10.1186/s40168-022-01320-0. PMID 35986393
- [Background] Galus L, Michalak M, Lorenz M, Stoinska-Swiniarek R, Tusien Malecka D, Galus A, Kolenda T, Leporowska E, Mackiewicz J. Vitamin D supplementation increases objective response rate and prolongs progression-free time in patients with advanced melanoma undergoing anti-PD-1 therapy. Cancer. 2023 Jul 1;129(13):2047-2055. doi: 10.1002/cncr.34718. Epub 2023 Apr 24. PMID 37089083
- [Background] Bosman ES, Albert AY, Lui H, Dutz JP, Vallance BA. Skin Exposure to Narrow Band Ultraviolet (UVB) Light Modulates the Human Intestinal Microbiome. Front Microbiol. 2019 Oct 24;10:2410. doi: 10.3389/fmicb.2019.02410. eCollection 2019. PMID 31708890
- [Background] Giampazolias E, Pereira da Costa M, Lam KC, Lim KHJ, Cardoso A, Piot C, Chakravarty P, Blasche S, Patel S, Biram A, Castro-Dopico T, Buck MD, Rodrigues RR, Poulsen GJ, Palma-Duran SA, Rogers NC, Koufaki MA, Minutti CM, Wang P, Vdovin A, Frederico B, Childs E, Lee S, Simpson B, Iseppon A, Omenetti S, Kelly G, Goldstone R, Nye E, Suarez-Bonnet A, Priestnall SL, MacRae JI, Zelenay S, Patil KR, Litchfield K, Lee JC, Jess T, Goldszmid RS, Reis e Sousa C. Vitamin D regulates microbiome-dependent cancer immunity. Science. 2024 Apr 26;384(6694):428-437. doi: 10.1126/science.adh7954. Epub 2024 Apr 25. PMID 38662827
- [Background] Di Modica M, Gargari G, Regondi V, Bonizzi A, Arioli S, Belmonte B, De Cecco L, Fasano E, Bianchi F, Bertolotti A, Tripodo C, Villani L, Corsi F, Guglielmetti S, Balsari A, Triulzi T, Tagliabue E. Gut Microbiota Condition the Therapeutic Efficacy of Trastuzumab in HER2-Positive Breast Cancer. Cancer Res. 2021 Apr 15;81(8):2195-2206. doi: 10.1158/0008-5472.CAN-20-1659. Epub 2021 Jan 22. PMID 33483370
- [Background] Gopalakrishnan V, Spencer CN, Nezi L, Reuben A, Andrews MC, Karpinets TV, Prieto PA, Vicente D, Hoffman K, Wei SC, Cogdill AP, Zhao L, Hudgens CW, Hutchinson DS, Manzo T, Petaccia de Macedo M, Cotechini T, Kumar T, Chen WS, Reddy SM, Szczepaniak Sloane R, Galloway-Pena J, Jiang H, Chen PL, Shpall EJ, Rezvani K, Alousi AM, Chemaly RF, Shelburne S, Vence LM, Okhuysen PC, Jensen VB, Swennes AG, McAllister F, Marcelo Riquelme Sanchez E, Zhang Y, Le Chatelier E, Zitvogel L, Pons N, Austin-Breneman JL, Haydu LE, Burton EM, Gardner JM, Sirmans E, Hu J, Lazar AJ, Tsujikawa T, Diab A, Tawbi H, Glitza IC, Hwu WJ, Patel SP, Woodman SE, Amaria RN, Davies MA, Gershenwald JE, Hwu P, Lee JE, Zhang J, Coussens LM, Cooper ZA, Futreal PA, Daniel CR, Ajami NJ, Petrosino JF, Tetzlaff MT, Sharma P, Allison JP, Jenq RR, Wargo JA. Gut microbiome modulates response to anti-PD-1 immunotherapy in melanoma patients. Science. 2018 Jan 5;359(6371):97-103. doi: 10.1126/science.aan4236. Epub 2017 Nov 2. PMID 29097493
- [Background] Hakozaki T, Richard C, Elkrief A, Hosomi Y, Benlaifaoui M, Mimpen I, Terrisse S, Derosa L, Zitvogel L, Routy B, Okuma Y. The Gut Microbiome Associates with Immune Checkpoint Inhibition Outcomes in Patients with Advanced Non-Small Cell Lung Cancer. Cancer Immunol Res. 2020 Oct;8(10):1243-1250. doi: 10.1158/2326-6066.CIR-20-0196. Epub 2020 Jul 27. PMID 32847937
- [Background] Jin Y, Dong H, Xia L, Yang Y, Zhu Y, Shen Y, Zheng H, Yao C, Wang Y, Lu S. The Diversity of Gut Microbiome is Associated With Favorable Responses to Anti-Programmed Death 1 Immunotherapy in Chinese Patients With NSCLC. J Thorac Oncol. 2019 Aug;14(8):1378-1389. doi: 10.1016/j.jtho.2019.04.007. Epub 2019 Apr 23. PMID 31026576
- [Background] Newsome RC, Gharaibeh RZ, Pierce CM, da Silva WV, Paul S, Hogue SR, Yu Q, Antonia S, Conejo-Garcia JR, Robinson LA, Jobin C. Interaction of bacterial genera associated with therapeutic response to immune checkpoint PD-1 blockade in a United States cohort. Genome Med. 2022 Mar 29;14(1):35. doi: 10.1186/s13073-022-01037-7. PMID 35346337
- [Background] Ren S, Feng L, Liu H, Mao Y, Yu Z. Gut microbiome affects the response to immunotherapy in non-small cell lung cancer. Thorac Cancer. 2024 May;15(14):1149-1163. doi: 10.1111/1759-7714.15303. Epub 2024 Apr 4. PMID 38572783
- [Background] Routy B, Le Chatelier E, Derosa L, Duong CPM, Alou MT, Daillere R, Fluckiger A, Messaoudene M, Rauber C, Roberti MP, Fidelle M, Flament C, Poirier-Colame V, Opolon P, Klein C, Iribarren K, Mondragon L, Jacquelot N, Qu B, Ferrere G, Clemenson C, Mezquita L, Masip JR, Naltet C, Brosseau S, Kaderbhai C, Richard C, Rizvi H, Levenez F, Galleron N, Quinquis B, Pons N, Ryffel B, Minard-Colin V, Gonin P, Soria JC, Deutsch E, Loriot Y, Ghiringhelli F, Zalcman G, Goldwasser F, Escudier B, Hellmann MD, Eggermont A, Raoult D, Albiges L, Kroemer G, Zitvogel L. Gut microbiome influences efficacy of PD-1-based immunotherapy against epithelial tumors. Science. 2018 Jan 5;359(6371):91-97. doi: 10.1126/science.aan3706. Epub 2017 Nov 2. PMID 29097494
- [Background] Salgia NJ, Bergerot PG, Maia MC, Dizman N, Hsu J, Gillece JD, Folkerts M, Reining L, Trent J, Highlander SK, Pal SK. Stool Microbiome Profiling of Patients with Metastatic Renal Cell Carcinoma Receiving Anti-PD-1 Immune Checkpoint Inhibitors. Eur Urol. 2020 Oct;78(4):498-502. doi: 10.1016/j.eururo.2020.07.011. Epub 2020 Aug 19. PMID 32828600
- [Background] Song P, Yang D, Wang H, Cui X, Si X, Zhang X, Zhang L. Relationship between intestinal flora structure and metabolite analysis and immunotherapy efficacy in Chinese NSCLC patients. Thorac Cancer. 2020 Jun;11(6):1621-1632. doi: 10.1111/1759-7714.13442. Epub 2020 Apr 23. PMID 32329229
- [Background] Tan J, McKenzie C, Potamitis M, Thorburn AN, Mackay CR, Macia L. The role of short-chain fatty acids in health and disease. Adv Immunol. 2014;121:91-119. doi: 10.1016/B978-0-12-800100-4.00003-9. PMID 24388214
- [Background] Zheng D, Liwinski T, Elinav E. Interaction between microbiota and immunity in health and disease. Cell Res. 2020 Jun;30(6):492-506. doi: 10.1038/s41422-020-0332-7. Epub 2020 May 20. PMID 32433595
- [Background] Barrea L, Muscogiuri G, Frias-Toral E, Laudisio D, Pugliese G, Castellucci B, Garcia-Velasquez E, Savastano S, Colao A. Nutrition and immune system: from the Mediterranean diet to dietary supplementary through the microbiota. Crit Rev Food Sci Nutr. 2021;61(18):3066-3090. doi: 10.1080/10408398.2020.1792826. Epub 2020 Jul 21. PMID 32691606
- [Background] Jannasch F, Kroger J, Schulze MB. Dietary Patterns and Type 2 Diabetes: A Systematic Literature Review and Meta-Analysis of Prospective Studies. J Nutr. 2017 Jun;147(6):1174-1182. doi: 10.3945/jn.116.242552. Epub 2017 Apr 19. PMID 28424256
- [Background] Sureda A, Bibiloni MDM, Julibert A, Bouzas C, Argelich E, Llompart I, Pons A, Tur JA. Adherence to the Mediterranean Diet and Inflammatory Markers. Nutrients. 2018 Jan 10;10(1):62. doi: 10.3390/nu10010062. PMID 29320413
- [Background] Covas MI, de la Torre R, Fito M. Virgin olive oil: a key food for cardiovascular risk protection. Br J Nutr. 2015 Apr;113 Suppl 2:S19-28. doi: 10.1017/S0007114515000136. PMID 26148918
- [Background] Meslier V, Laiola M, Roager HM, De Filippis F, Roume H, Quinquis B, Giacco R, Mennella I, Ferracane R, Pons N, Pasolli E, Rivellese A, Dragsted LO, Vitaglione P, Ehrlich SD, Ercolini D. Mediterranean diet intervention in overweight and obese subjects lowers plasma cholesterol and causes changes in the gut microbiome and metabolome independently of energy intake. Gut. 2020 Jul;69(7):1258-1268. doi: 10.1136/gutjnl-2019-320438. Epub 2020 Feb 19. PMID 32075887
- [Background] Morze J, Danielewicz A, Przybylowicz K, Zeng H, Hoffmann G, Schwingshackl L. An updated systematic review and meta-analysis on adherence to mediterranean diet and risk of cancer. Eur J Nutr. 2021 Apr;60(3):1561-1586. doi: 10.1007/s00394-020-02346-6. Epub 2020 Aug 8. PMID 32770356
- [Background] Castro-Espin C, Bonet C, Crous-Bou M, Nadal-Zaragoza N, Tjonneland A, Mellemkjaer L, Hajji-Louati M, Truong T, Katzke V, Le Cornet C, Schulze MB, Jannasch F, Masala G, Sieri S, Panico S, Di Girolamo C, Skeie G, Borch KB, Olsen KS, Sanchez MJ, Amiano P, Chirlaque MD, Guevara M, Sund M, Boden S, Gunter MJ, Gonzalez-Gil EM, Weiderpass E, Aguilera-Buenosvinos I, Tsilidis KK, Heath AK, Aune D, Dossus L, Agudo A. Association of Mediterranean diet with survival after breast cancer diagnosis in women from nine European countries: results from the EPIC cohort study. BMC Med. 2023 Jun 26;21(1):225. doi: 10.1186/s12916-023-02934-3. PMID 37365585
- [Background] Buckland G, Travier N, Cottet V, Gonzalez CA, Lujan-Barroso L, Agudo A, Trichopoulou A, Lagiou P, Trichopoulos D, Peeters PH, May A, Bueno-de-Mesquita HB, Bvan Duijnhoven FJ, Key TJ, Allen N, Khaw KT, Wareham N, Romieu I, McCormack V, Boutron-Ruault M, Clavel-Chapelon F, Panico S, Agnoli C, Palli D, Tumino R, Vineis P, Amiano P, Barricarte A, Rodriguez L, Sanchez MJ, Chirlaque MD, Kaaks R, Teucher B, Boeing H, Bergmann MM, Overvad K, Dahm CC, Tjonneland A, Olsen A, Manjer J, Wirfalt E, Hallmans G, Johansson I, Lund E, Hjartaker A, Skeie G, Vergnaud AC, Norat T, Romaguera D, Riboli E. Adherence to the mediterranean diet and risk of breast cancer in the European prospective investigation into cancer and nutrition cohort study. Int J Cancer. 2013 Jun 15;132(12):2918-27. doi: 10.1002/ijc.27958. Epub 2012 Dec 19. PMID 23180513
- [Background] McHugh A, O'Connell E, Gurd B, Rae P, George ES, Kleckner AS, Baguley BJ. Mediterranean-style dietary interventions in adults with cancer: a systematic review of the methodological approaches, feasibility, and preliminary efficacy. Eur J Clin Nutr. 2024 Jun;78(6):463-476. doi: 10.1038/s41430-024-01426-8. Epub 2024 Mar 8. PMID 38459161
- [Background] Ahmad S, Moorthy MV, Lee IM, Ridker PM, Manson JE, Buring JE, Demler OV, Mora S. Mediterranean Diet Adherence and Risk of All-Cause Mortality in Women. JAMA Netw Open. 2024 May 1;7(5):e2414322. doi: 10.1001/jamanetworkopen.2024.14322. PMID 38819819
- [Background] Harvey BI, Youngblood SM, Kleckner AS. Barriers and Facilitators to Adherence to a Mediterranean Diet Intervention during Chemotherapy Treatment: A Qualitative Analysis. Nutr Cancer. 2023;75(5):1349-1360. doi: 10.1080/01635581.2023.2192891. Epub 2023 Mar 20. PMID 36942399
- [Background] Kiani AK, Medori MC, Bonetti G, Aquilanti B, Velluti V, Matera G, Iaconelli A, Stuppia L, Connelly ST, Herbst KL, Bertelli M. Modern vision of the Mediterranean diet. J Prev Med Hyg. 2022 Oct 17;63(2 Suppl 3):E36-E43. doi: 10.15167/2421-4248/jpmh2022.63.2S3.2745. eCollection 2022 Jun. PMID 36479477
- [Background] Hanahan D. Hallmarks of Cancer: New Dimensions. Cancer Discov. 2022 Jan;12(1):31-46. doi: 10.1158/2159-8290.CD-21-1059. PMID 35022204
- [Background] Sender R, Fuchs S, Milo R. Revised Estimates for the Number of Human and Bacteria Cells in the Body. PLoS Biol. 2016 Aug 19;14(8):e1002533. doi: 10.1371/journal.pbio.1002533. eCollection 2016 Aug. PMID 27541692
- [Background] Exarchakou A, Kipourou DK, Belot A, Rachet B. Socio-economic inequalities in cancer survival: how do they translate into Number of Life-Years Lost? Br J Cancer. 2022 Jun;126(10):1490-1498. doi: 10.1038/s41416-022-01720-x. Epub 2022 Feb 11. PMID 35149855
- [Background] Vaccarella S, Lortet-Tieulent J, Saracci R, Fidler MM, Conway DI, Vilahur N, Sarfati D, Jemal A, Mackenbach JP, Marmot MG, Straif K, Wild CP. Reducing Social Inequalities in Cancer: Setting Priorities for Research. CA Cancer J Clin. 2018 Sep;68(5):324-326. doi: 10.3322/caac.21463. Epub 2018 Jul 10. No abstract available. PMID 30152865
- [Background] Dalton SO, Olsen MH, Johansen C, Olsen JH, Andersen KK. Socioeconomic inequality in cancer survival - changes over time. A population-based study, Denmark, 1987-2013. Acta Oncol. 2019 May;58(5):737-744. doi: 10.1080/0284186X.2019.1566772. Epub 2019 Feb 11. PMID 30741062
- [Background] Lundqvist A, Andersson E, Ahlberg I, Nilbert M, Gerdtham U. Socioeconomic inequalities in breast cancer incidence and mortality in Europe-a systematic review and meta-analysis. Eur J Public Health. 2016 Oct;26(5):804-813. doi: 10.1093/eurpub/ckw070. Epub 2016 May 23. PMID 27221607
- [Background] Vaccarella S, Lortet-Tieulent J, Saracci R, Conway DI, Straif K, Wild CP, editors. Reducing social inequalities in cancer: evidence and priorities for research. Lyon (FR): International Agency for Research on Cancer; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK566181/ PMID 33443989
- [Background] Hurria A, Jones L, Muss HB. Cancer Treatment as an Accelerated Aging Process: Assessment, Biomarkers, and Interventions. Am Soc Clin Oncol Educ Book. 2016;35:e516-22. doi: 10.1200/EDBK_156160. PMID 27249761
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Long-term outcomes for neoadjuvant versus adjuvant chemotherapy in early breast cancer: meta-analysis of individual patient data from ten randomised trials. Lancet Oncol. 2018 Jan;19(1):27-39. doi: 10.1016/S1470-2045(17)30777-5. Epub 2017 Dec 11. PMID 29242041
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Gamrath L, Pedersen TB, Moller MV, Volmer LM, Holst-Christensen L, Vestermark LW, Donskov F. Role of the Microbiome and Diet for Response to Cancer Checkpoint Immunotherapy: A Narrative Review of Clinical Trials. Curr Oncol Rep. 2025 Jan;27(1):45-58. doi: 10.1007/s11912-024-01622-6. Epub 2025 Jan 3. PMID 39753816
- See also: Nordic registry of cancer incidences and mortality — https://nordcan.iarc.fr/